CLINICAL TRIAL: NCT06644404
Title: A Randomized, Open, Two-sequence, Crossover, Multiple Oral Administrations, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Drug-drug Interaction Between DWP16001, DWC202407, and DWC202408 in Healthy Adults
Brief Title: Phase 1 Study of Drug-Drug Interactions Between DWP16001, DWC202407, and DWC202408 in Healthy Adults
Acronym: DW_DWP16001112
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001112
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enavogliflozin 0.3mg, once daily (Experimental)
  Interventions: Drug: DWP16001 0.3mg
- Metformin 1,000mg, BID (Experimental)
  Interventions: Drug: DWC202407 1,000mg
- Glimepiride 2mg, once daily (Experimental)
  Interventions: Drug: DWC202408 2mg

INTERVENTIONS:
Drug: DWP16001 0.3mg — 1 tablet, Orally, Once daily single dose
  Arms: Enavogliflozin 0.3mg, once daily
Drug: DWC202407 1,000mg — 1 tablet, Orally, Twice daily
  Arms: Metformin 1,000mg, BID
Drug: DWC202408 2mg — 1 tablet, Orally, Once daily single dose
  Arms: Glimepiride 2mg, once daily

SUMMARY:
This study aims to evaluate the pharmacokinetic/pharmacodynamic drug-drug interactions between DWP16001, DWC202407, and DWC202408 in healthy adults

DETAILED DESCRIPTION:
This study aims to evaluate the pharmacokinetic interactions, pharmacodynamic interactions, safety, and tolerability of DWP16001, DWC202407, and DWC202408 in healthy adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged 19 to 50 years at the time of screening.
2. Individuals with a body weight between 50.0 kg and 90.0 kg and a Body Mass Index (BMI) between 18.5 kg/m² and 29.9 kg/m² at the time of screening.
3. Female volunteers must be neither pregnant nor breastfeeding, or must be in a surgically sterile state (e.g., bilateral tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy).
4. Individuals who have been fully informed about the clinical trial, have fully understood the details, voluntarily decided to participate, and provided written consent to comply with the precautions.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10-26 (Estimated); Primary Completion 2024-12-03 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss of DWP16001 | 0-24 hours
  Peak Plasma Concentration at steady-state
AUCtau,ss of DWP16001 | 0-24 hours
  Area under the plasma concentration versus time curve at Tau, steady-state
Cmax,ss of DWC202407 | 0-12 hours
  Peak Plasma Concentration at steady-state
AUCtau,ss of DWC202407 | 0-12 hours
  Area under the plasma concentration versus time curve at Tau, steady-state
Cmax,ss of DWC202408 | 0-24 hours
  Peak Plasma Concentration at steady-state
AUCtau,ss of DWC202408 | 0-24 hours
  Area under the plasma concentration versus time curve at Tau, steady-state

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No